CLINICAL TRIAL: NCT02909764
Title: Salty Taste: Assessing a Strategy to Reduce Children's Preference
Brief Title: Shifting Salty Taste Preferences in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Monell Chemical Senses Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 823281
Record Dates: First submitted 2016-09-01; First posted 2016-09-21 (Estimated); Results first posted 2019-08-20 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Development
Keywords: Salty taste; Psychophysics; Genetics; Diet; Age

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Children will receive regularly salted cereal to consume 4 times per week over a 2-month period.
- Low Sodium Group (Experimental): Intervention: Children will receive low sodium cereal to consume 4 times per week over a 2-month period.
  Interventions: Other: Low Sodium Group

INTERVENTIONS:
Other: Low Sodium Group — Breakfast Cereal
  Arms: Low Sodium Group

SUMMARY:
The goals of the proposed research are to determine whether repeated exposure to a low sodium food will result in reduced preference for salt in that food among children; and to determine whether such reductions in preference are related to dietary intake of salt, taste receptor genotype, and anthropometric and physiological measures.

DETAILED DESCRIPTION:
This is a within- and between-subjects randomized controlled trial on children consuming either a low sodium or a higher sodium cereal over a 2-month period to determine if repeated exposure to the low sodium cereal is effective for reducing preference for salt in that food. Children will be genotyped for markers related to taste, dietary intake will be recorded, and anthropometric and physiological measures will be collected at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Willingness to consume no other cereals during intervention

Exclusion Criteria:

* Allergies and/or taking medication that affects taste

Ages: 7 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Mennella, PhD, Principal Investigator — Monell Chemical Senses Center
Locations (1):
- Monell Chemical Senses Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bobowski N, Mennella JA. Repeated Exposure to Low-Sodium Cereal Affects Acceptance but Does not Shift Taste Preferences or Detection Thresholds of Children in a Randomized Clinical Trial. J Nutr. 2019 May 1;149(5):870-876. doi: 10.1093/jn/nxz014. PMID 31006818

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Mothers were recruited from a list of past participants in our research program who asked to be contacted for future studies. Study was conducted at The Monell Chemical Senses Center in Philadelphia, Pennsylvania USA in 2016.
Pre-assignment Details: Children were randomized at the beginning of the first test session. There were no significant effects that occurred after participant enrollment but before randomization to study group.
Groups:
- Control Group [Regular Sodium Group]: Children will receive regularly salted cereal to consume 4 times per week over an 8-week (2-month) period.
- Low Sodium Group: Intervention: Children will receive low sodium cereal to consume 4 times per week over an 8-week (2-month) period.
  Low Sodium Group: Breakfast Cereal
Period: Overall Study
Arm/Group | Control Group [Regular Sodium Group] | Low Sodium Group
Started | 19 | 20
Completed | 19 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control Group [Regular Sodium Group]: Children will receive regularly salted cereal to consume 4 times per week over a 2-month period.
- Total: Total of all reporting groups
Arm/Group | Control Group [Regular Sodium Group] | Low Sodium Group | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.4 (2.3) | 11.3 (2.2) | 11.3 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 6 | 7 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 16 | 26
  White | 3 | 2 | 5
  More than one race | 6 | 2 | 8
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Most Preferred Level of Salt Taste
Description: Children were presented with pairs of broths with varying concentrations of added salt (0.16, 0.24, 0.38, 0.61, 1.05 M) (17) . The first pair of broths (0.24 and 0.61 M salt) presented were from the middle range of concentrations. Children were instructed to taste each sample within a pair for 5 seconds, to rinse between tastings, and then to point to the sample they liked better. Each subsequent pair of samples contained the concentration selected by the participant paired with an adjacent stimulus concentration. This pattern continued until the child either chose the same concentration when paired with both a lower and higher concentration in two consecutive pairs or chose either the highest or the lowest concentration twice consecutively. The entire task was repeated a, with stimulus pairs presented in reverse order. The geometric mean of the two concentrations chosen in the first and second series was calculated to determine most preferred levels of salt.
Time Frame: Baseline (time 0) and after 8-week intervention
Population: Some children did not understand the task and responded at random.
Measure: Geometric Mean (Standard Error); unit: mol/L
Arm/Group | Control Group [Regular Sodium Group] | Low Sodium Group
Number analyzed (Participants) | 19 | 20
mol/L
  Baseline: number analyzed (Participants) | 16 | 16
  Baseline | 0.44 (0.04) | 0.34 (0.04)
  After 8-week intervention: number analyzed (Participants) | 16 | 16
  After 8-week intervention | 0.42 (0.05) | 0.43 (0.05)
Statistical Analysis 1: Comparison: Control Group [Regular Sodium Group] vs Low Sodium Group; Test type: Other; p = 0.30, ANOVA

2. Primary Outcome: Relative Preference for Regular vs Low Sodium Cereal
Description: The number of children who preferred the taste of the low salt cereal when compared to the regular sodium cereal
Time Frame: At baseline and after 8-week intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group [Regular Sodium Group] | Low Sodium Group
Number analyzed (Participants) | 19 | 20
Participants
  Baseline, Number preferred low salt cereal | 3 | 5
  End Intervention, Number preferred low salt cereal | 7 | 4
Statistical Analysis 1: Comparison: Control Group [Regular Sodium Group] vs Low Sodium Group; Yates's chi-square analyses were used to determine which of the two cereals children in each group preferred at baseline and after the 8-week exposure period, and whether the number of children who shifted preference from the regular cereal at baseline to the low salt cereal after the exposure period differed between groups; Test type: Other — Yates's chi-square analyses were used to determine which of the two cereals children in each group preferred at baseline and after the 8-week exposure period, and whether the number of children who shifted preference from the regular cereal at baseline to the low salt cereal after the exposure period differed between groups; p < 0.05, Chi-squared

3. Secondary Outcome: Salt Taste Detection Thresholds
Description: Detection thresholds (the lowest level of salt detect by taste) were measured via a two-alternative forced-choice procedure
Time Frame: Baseline and after 8-week intervention
Population: Some children did not understand or complete the task.
Measure: Mean (Standard Error); unit: mol x 10-3/L
Arm/Group | Control Group [Regular Sodium Group] | Low Sodium Group
Number analyzed (Participants) | 19 | 20
mol x 10-3/L
  Baseline: number analyzed (Participants) | 16 | 15
  Baseline | 4.4 (0.8) | 3.6 (0.8)
  After 8-week Exposure Period: number analyzed (Participants) | 16 | 15
  After 8-week Exposure Period | 4.6 (1.0) | 5.4 (1.1)
Statistical Analysis 1: Comparison: Control Group [Regular Sodium Group] vs Low Sodium Group; Test type: Other; p = 0.32, ANOVA

4. Secondary Outcome: Most Preferred Level of Sucrose
Description: Children were presented with pairs of sucrose solutions of varying concentrations (0.09, 0.18, 0.35, 0.70, 1.05 M). The first pair presented were from the middle range of concentrations. Children tasted each sample and then pointed to the sample they liked better. Each subsequent pair of samples presented contained the concentration selected by the child paired with an adjacent stimulus concentration. This pattern continued until the child either chose the same concentration when paired with both a lower and higher concentration in two consecutive pairs or chose either the highest or the lowest concentration twice consecutively. The entire task was repeated after a 3-minute break, with stimulus pairs presented in reverse order. The geometric mean of the two concentrations chosen in the first and second series was calculated to determine the most preferred levels of sucrose.
Time Frame: At baseline and after 8-week intervention
Measure: Geometric Mean (Standard Error); unit: mol/L
Arm/Group | Control Group [Regular Sodium Group] | Low Sodium Group
Number analyzed (Participants) | 19 | 20
mol/L
  Baseline | 0.72 (0.07) | 0.57 (0.07)
  After 8-week intervention | 0.76 (0.06) | 0.64 (0.06)
Statistical Analysis 1: Comparison: Control Group [Regular Sodium Group] vs Low Sodium Group; Test type: Other; p = 0.77, ANOVA

5. Secondary Outcome: Intake of Cereal During Intervention Period
Description: Mothers recorded the amount of cereal their children ingested during 28 days of the 8-week, at-home intervention period.
Time Frame: 28 days
Measure: Mean (Standard Error); unit: grams
Arm/Group | Control Group [Regular Sodium Group] | Low Sodium Group
Number analyzed (Participants) | 19 | 20
grams
  Intake, Day 1 | 27.8 (4.3) | 19.3 (4.7)
  Intake, Day 2 | 33.3 (4.3) | 17.9 (4.7)
  Intake, Day 3 | 30.6 (4.3) | 18.9 (4.7)
  Intake, Day 4 | 34.8 (4.3) | 19.8 (4.7)
  Intake, Day 5 | 25.7 (4.3) | 20.3 (4.7)
  Intake, Day 6 | 27.8 (4.3) | 19.4 (4.7)
  Intake, Day 7 | 27.0 (4.3) | 20.3 (4.7)
  Intake, Day 8 | 24.9 (4.3) | 19.3 (4.7)
  Intake, Day 9 | 24.9 (4.3) | 16.5 (4.7)
  Intake, Day 10 | 23.4 (4.3) | 17.6 (4.7)
  Intake, Day 11 | 25.9 (4.3) | 16.5 (4.7)
  Intake, Day 12 | 24.5 (4.3) | 15.3 (4.7)
  Intake, Day 13 | 24.5 (4.3) | 17.7 (4.9)
  Intake, Day 14 | 24.9 (4.3) | 15.4 (4.9)
  Intake, Day 15 | 24.2 (4.4) | 19.4 (4.9)
  Intake, Day 16 | 23.2 (4.4) | 18.9 (5.0)
  Intake, Day 17 | 24.2 (4.7) | 13.9 (5.2)
  Intake, Day 18 | 27.0 (4.7) | 15.7 (5.2)
  Intake, Day 19 | 23.7 (4.7) | 12.6 (5.2)
  Intake, Day 20 | 21.8 (4.7) | 14.3 (5.2)
  Intake, Day 21 | 20.2 (4.7) | 16.4 (5.2)
  Intake, Day 22 | 25.9 (4.7) | 15.7 (5.2)
  Intake, Day 23 | 23.8 (4.7) | 12.5 (5.2)
  Intake, Day 24 | 23.0 (4.7) | 11.3 (5.2)
  Intake, Day 25 | 25.8 (4.7) | 15.7 (5.2)
  Intake, Day 26 | 23.5 (4.7) | 13.7 (5.2)
  Intake, Day 27 | 19.0 (4.7) | 12.5 (5.2)
  Intake, Day 28 | 23.0 (4.7) | 10.7 (5.2)
Statistical Analysis 1: Comparison: Control Group [Regular Sodium Group] vs Low Sodium Group; Generalized estimating equations (GEE) were conducted on the amount of cereal in grams ingested during 28 days home-exposure period. The GEE approach accounts for the repeated measurements of outcomes over time for each child and examines whether the slopes of the lines created differ between the treatment groups; Test type: Other — General estimating equations (GEE); p < 0.05, GEE

6. Secondary Outcome: Blood Pressure
Description: Blood pressure (mmHg) was measured by using an automatic blood pressure machine with pediatric cuff. Blood pressure will be measured at baseline (time 0). There were no a priori hypothesis but were collected as baseline characteristic to ensure no differences between the groups.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Control Group | Low Sodium Group
Number analyzed (Participants) | 18 | 20
mmHg
  Systolic, baseline | 113.7 (2.7) | 115.5 (2.9)
  Diastolic, baseline | 65.1 (1.3) | 66.6 (1.4)
Statistical Analysis 1: Comparison: Control Group vs Low Sodium Group; T-tests were conducted to determine whether differences in baseline blood pressure between the two groups; Test type: Other — T-tests were conducted to determine whether differences in baseline blood pressure between groups; p > 0.40, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 4 month
Arm/Group | Control Group [Regular Sodium Group] | Low Sodium Group
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 0/19 | 0/20

LIMITATIONS AND CAVEATS:
We did not collect reliable diet records so no data were available to report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No